CLINICAL TRIAL: NCT00791375
Title: Web-based Physical Activity Intervention for Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Carolyn Rabin, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CA134197; 1R03CA134197 (NIH)
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Cancer
Keywords: young adult; cancer; exercise; physical activity
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity Intervention (Experimental): Participants in this arm will be given access to a website designed to help them increase their levels of physical activity
  Interventions: Behavioral: Physical activity intervention
- Cancer Website Control Group (Placebo Comparator): Participants in this arm will be given information on cancer-related websites (that do not provide information on physical activity)
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention — Comparison of providing access to a targeted physical activity web-site v. providing information on cancer-related websites

SUMMARY:
The goal of this study is to adapt a previously developed web-based physical activity intervention so that the intervention targets young adult cancer survivors(age 18 to 39). The web-based intervention will then be pilot tested to determine whether it is feasible for and acceptable to young adult cancer survivors; we hypothesize that the intervention will be both feasible and acceptable. Preliminary data on the effects of the intervention on physical activity level, mood and fatigue will also be collected.

DETAILED DESCRIPTION:
Young adults diagnosed with cancer constitute a particularly vulnerable population whose medical and psychosocial needs are often overlooked. Those diagnosed with cancer between the ages of 18 and 39 face a number of increased risks including an increased risk of cardiovascular disease, second cancers, and emotional distress. Despite this, only a very small percentage of cancer research has focused on the survivorship issues of young adults. The goal of the proposed research is to address some of the unmet needs among young adult cancer survivors by developing and pilot testing a physical activity intervention for this population. Physical activity was selected as the target behavior as: 1. a high percentage of young adult cancer survivors have a sedentary lifestyle and 2. research has shown that cancer survivors who increase their physical activity experience improved cardiopulmonary function, reduced fatigue, enhanced mood and superior cancer outcomes. The intervention will be based on a previously developed, theoretically-grounded, tailored Internet intervention for sedentary adults. This previously developed intervention uses components of the Transtheoretical Model and Social Cognitive Theory to promote physical activity; for example, participants complete monthly questionnaires online and received tailored feedback reports addressing their self-efficacy, decisional balance and processes of change. The intervention website also includes features such as tips for exercising while caring for young children and local physical activity resources. Two key enhancements will be added to the intervention website in order to target the young adult cancer survivor population- 1. information pertinent to cancer survivors initiating an exercise program and 2. a peer-to-peer support component. Once these enhancements have been added, 10 young adult cancer survivors will evaluate the intervention and provide qualitative feedback. Additional revisions will be made to the intervention, as needed, based on this feedback. The intervention will then be pilot tested with a sample of 40 young adult cancer survivors. Participants will be randomly assigned to an intervention group (receiving 12 weeks of access to the intervention website) or a comparison group (receiving information on three cancer-specific Internet sites). Data on intervention feasibility and acceptability will be collected along with preliminary data on intervention effects (i.e., on physical activity level, mood, and fatigue). The latter will be used for effect size estimates when designing a future efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 39
* diagnosed with any form of cancer (except non-melanoma skin cancer) between the ages of 18 and 39 in the past 10 years
* completed all surgery, chemotherapy and radiation therapy
* currently in a cancer remission
* able to speak and write fluently in English
* able to access the Internet (at home, school, or work)
* sedentary.

Exclusion Criteria:

* currently pregnant or the intention to get pregnant
* the presence of a known medical condition (e.g., history of CVD) or history of severe psychiatric illness (e.g., psychotic disorder) making participation dangerous or very difficult

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Feasibility measure: percentage of weeks that participants enter physical activity goals and information on the intervention website | 12 weeks
Acceptability measure: response to the item "In general how satisfied were you with the intervention?" | 12 weeks

SECONDARY OUTCOMES:
Minutes of moderate-intensity activity on Seven Day PAR | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Rabin, Principal Investigator — The Miriam Hospital
Locations (1):
- Miriam Hospital, Providence, Rhode Island, United States